CLINICAL TRIAL: NCT06195072
Title: Platform Clinical Study for Conquering Scleroderma: A Multicenter, Double-Blind, Randomized, Placebo-Controlled, Phase 2b Platform Clinical Study to Evaluate the Safety and Efficacy of Investigational Products in Participants With Interstitial Lung Disease Secondary to Systemic Sclerosis
Brief Title: Platform Clinical Study for Conquering Scleroderma
Acronym: CONQUEST
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Scleroderma Research Foundation, Inc. (Other)
Collaborators: Sanofi (Industry); Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SRF201
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-10

CONDITIONS: Interstitial Lung Disease Due to Systemic Disease; Scleroderma
Keywords: platform; scleroderma; interstitial lung disease; systemic sclerosis; SSc; SSc-ILD
MeSH Terms: conditions — Scleroderma, Diffuse; Lung Diseases, Interstitial; Scleroderma, Systemic | interventions — BI 1015550

STUDY DESIGN:
Intervention Model Description: Participants who have given informed consent for the Master Protocol and all available Regimen-specific Subprotocols for which they are eligible will be randomly assigned to a regimen. Within each regimen, participants will be assigned to active treatment or matching placebo in a ratio detailed in the randomization scheme.
  Eligibility for the Regimen will be based on the inclusion and exclusion criteria in the Master Protocol and on the inclusion and exclusion criteria in the Regimen-specific Subprotocol.
  Importantly, to preserve the integrity of randomization, participants will be consented to all possible Regimen-specific Subprotocols open at that time, for which they qualify. Eligible participants will then be randomized to only one Regimen-specific Subprotocol, followed by randomization to the active IP treatment or to the corresponding placebo within a Regimen-specific Subprotocol.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: There will be multiple interventional regimens, each consisting of the study participants receiving either the active IP or its matching placebo. Study participants, Investigators, and site staff will not be blinded to the regimen assignment, but they will be blinded to active product or matching placebo assignment. Enrollment to regimens may start at different time points during the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Amlitelimab (Experimental)
  Interventions: Drug: Amlitelimab
- Amlitelimab matching placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- BI 1015550 (Nerandomilast) (Experimental)
  Interventions: Drug: BI 1015550 (Nerandomilast)
- BI 1015550 (Nerandomilast) matching placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amlitelimab — IP will be administered subcutaneously by the Investigator or designee as follows:
  * Amlitelimab or
  * Matching placebo
  Arms: Amlitelimab
Drug: BI 1015550 (Nerandomilast) — Study participants will take the active investigational product BI 1015550 (Nerandomilast) or matching placebo provided as film-coated tablets, administered orally BID.
  Arms: BI 1015550 (Nerandomilast)
Drug: Placebo — see Experimental Arm intervention description
  Arms: Amlitelimab matching placebo; BI 1015550 (Nerandomilast) matching placebo

SUMMARY:
The goal of this clinical trial is to test efficacy of different investigational products (IPs) compared with placebo on the change from baseline to the end of the treatment period at Week 52 in lung capacity in participants with Interstitial Lung Disease Secondary to Systemic Sclerosis.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18+ years of age at the time of signed informed consent;
2. SSc classification as defined by the 2013 American College of Rheumatology/European League Against Rheumatism criteria. Participants with diffuse, limited or sine cutaneous skin involvement are eligible
3. Onset of SSc (defined by first non-Raynaud's symptom) 7 years or less prior to the Screening Visit;
4. A Modified Rodnan skin score (mRSS) less than 40
5. Presence of ILD with evidence of any fibrosis on HRCT (within 3 months or less of randomization)
6. Presence of an FVC 45% or more predicted normal;
7. Presence of a diffusing capacity of the lung for carbon monoxide (DLCO) 30% or more predicted normal, corrected for hemoglobin;

Other protocol and/or subprotocol inclusion criteria apply.

Exclusion Criteria:

1. Presence of clinically significant pulmonary abnormalities inconsistent with ILD on HRCT (e.g., scarring due to previous active tuberculosis [TB], sarcoidosis, lung mass, or other findings unrelated to SSc-ILD, as determined by a local radiologist/Investigator);
2. Presence of infected ulcers or active gangrene at the Screening Visit;
3. History of scleroderma renal crisis within 6 months prior to the Screening Visit;
4. Forced expiratory volume in 1 second/FVC <0.65 (pre-bronchodilator) at the Screening Visit
5. History of stem cell transplantation, bone marrow transplantation, chimeric antigen receptor T-cell therapy, or solid organ transplantation;
6. History of treatment with rituximab within the 6 months prior to the Screening Visit;
7. History treatment with cell-depleting therapies other than rituximab, including, but not limited to, CAMPATH®; anti-cluster of differentiation (CD)3, anti-CD4, anti-CD5, antiCD19, and anti-CD20 agents; and investigational agents
8. Treatment with tocilizumab, nintedanib, pirfenidone, abatacept, leflunomide, tacrolimus, tofacitinib, intravenous immunoglobulin (IVIG), or any biologic or cyclophosphamide within 3 months prior to Screening Visit
9. History of use of any investigational medication or device for any indication within 30 days or 5 half-lives (whichever is longer) prior to Screening Visit.
10. Presence of any of the following laboratory findings at the Screening Visit:

    * Estimated glomerular filtration rate <45 mL/min/1.73 m2, calculated using the Chronic Kidney Disease Epidemiology Collaboration equation;
    * Alanine aminotransferase or aspartate aminotransferase level > (2 x ULN);
    * Platelets <100 × 109/L (100,000/μL);
    * White blood cell count <2500/μL;
    * Neutrophil blood count <1500/μL;
    * Prothrombin time and partial thromboplastin time >1.5 × ULN, or international normalized ratio >2; or
    * Any other laboratory test result, that in the opinion of the Investigator, might place the study participant at risk for participation in the study.
11. Presence of a clinically significant disorder that, in the opinion of the Investigator, could contraindicate the administration of study product, affect compliance, interfere with study evaluations, or confound the interpretation of study results
12. Presence of a concomitant life-threatening disease with life expectancy <12 months based on the Investigator's assessment;
13. Evidence of active tuberculosis (TB) or being at high risk for TB

Other protocol and/or subprotocol exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
The change in forced vital capacity (FVC, in mL). | from baseline to the end of the treatment period at Week 52

SECONDARY OUTCOMES:
The percent change in high-resolution computed tomography (HRCT) quantitative interstitial lung disease - whole lung (QILD-WL); | from baseline to the end of the treatment period at Week 52
  Lung involvement as measured by high-resolution computed tomography (HRCT) assessed by quantitative interstitial lung disease - whole lung (QILD-WL)
The change in Functional Assessment of Chronic Illness Therapy (FACIT)-Dyspnea score. | from baseline to the end of the treatment period at Week 52
  Dyspnea (severity and functional limitations) are measured by the Functional Assessment of Chronic Illness Therapy (FACIT) - Dyspnea score. Dyspnea score range 0-4, total score 0-30 (higher score = worse outcome).
The proportion of study participants with an improvement in the revised CRISS score, in study participants with diffuse cutaneous SSc and baseline mRRS ≥10. | baseline, Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Kevin O'Shea, Study Chair — Scleroderma Research Foundation
Locations (34):
- United States (34):
  - University of Alabama - Division of Pulmonary and Critical Care Medicine, Birmingham, Alabama
  - Keck School of Medicine at USC Medical Center, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California, Los Angeles (UCLA) Ronald Reagan Medical Center, Los Angeles, California
  - Stanford University Medical Center, Palo Alto, California
  - Yale University School of Medicine - Epilepsy, New Haven, Connecticut
  - Georgetown University Medical Center - Department of Rheumatology, Washington D.C., District of Columbia
  - Emory University School of Medicine, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - The University of Chicago Medical Center (UCMC), Chicago, Illinois
  - University of Kansas School of Medicine, Kansas City, Kansas
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston University (BU), Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Northwell Health, Great Neck, New York
  - Hospital for Special Surgery, New York, New York
  - Columbia University Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health & Science University (OHSU), Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Meharry Medical College, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Houston - Division of Rheumatology and Clinical Immunogenetics, Houston, Texas
  - The University of Utah Health Sciences Center, Salt Lake City, Utah
  - Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khanna D, Evnin LB, Assassi S, Benton WW, Gordon G, Maslova K, Steffgen J, Maher TM. Design of CONQUEST, a novel, randomized, placebo-controlled, Phase 2b platform clinical trial to investigate new treatments for patients with early active systemic sclerosis with interstitial lung disease. J Scleroderma Relat Disord. 2024 Nov 5;10(2):121-132. doi: 10.1177/23971983241278079. eCollection 2025 Jun. PMID 39544897